CLINICAL TRIAL: NCT02868463
Title: Bladder Environment: Microbiome Oxygen Relationship
Acronym: BEMOR
Status: Completed | Type: Observational
Sponsor: Loyola University (Other)
Collaborators: Alan J. Wolfe (Unknown)
Responsible Party: Principal Investigator, Elizabeth Mueller, MD, Professor, Loyola University
Other Study IDs: 208221
Record Dates: First submitted 2016-08-04; First posted 2016-08-16 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Urinary Incontinence; UTI's
Keywords: oxygen tension; Female Urinary Microbiome; Urinary Tract Symptoms; Urine Oxygen Level
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine samples will be frozen and stored in the event additional analysis is necessary
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize bladder urinary oxygen tension (BUOT) in women whose urinary microbiomes contains at least one anaerobic bacterial species versus women whose urinary microbiomes do not contain anaerobes.

DETAILED DESCRIPTION:
Throughout the human body, microbial communities (microbiota) depend on their environment, including the level of oxygen (anaerobic vs. aerobic). Recently published evidence documents the existence of a female urinary microbiota (FUM) and provides evidence that the FUM differ based on lower urinary tract symptoms, i.e. no bladder symptoms, urgency urinary incontinence, and urinary tract infection1-4. Members of the FUM include bacteria that require oxygen (aerobes), those that abhor oxygen (anaerobes) and those that thrive in both conditions (facultative anaerobes)5. This last group of microbes is known to consume low levels of oxygen to maintain an anaerobic environment. Yet, virtually nothing is known about oxygen levels in bladder urine even though bladder urine oxygen tension may both affect and be affected by the FUM. Given the role oxygen levels play in other parts of the human body, the investigators request resources to investigate bladder urine oxygen levels. The study is designed to understand if BUOT levels differ in FUMs with and without at least one anaerobe, and if so, if there are any patient factors or urinary symptoms associated with certain BUOT

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* No indwelling urethral catheter
* At least 50 mL of urine in their bladder as determined by the clinic's bladder scanner

Exclusion Criteria:

* Non-English speaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female only participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Oxygen Tension Measurement of Bladder Urine and Correlation of These Oxygen Profiles with Expanded Urine Culture Bacterial Growth in Women | The study completion is expected at 2 years.
  Throughout the human body, microbial communities (microbiota) depend on their environment, including the level of oxygen (anaerobic vs. aerobic). Recently published evidence documents the existence of a female urinary microbiota (FUM) and provides evidence that the FUM differ based on lower urinary tract symptoms, i.e. no bladder symptoms, urgency urinary incontinence, and urinary tract infection. Members of the FUM include bacteria that require oxygen (aerobes), those that abhor oxygen (anaerobes) and those that thrive in both conditions (facultative anaerobes). This last group of microbes is known to consume low levels of oxygen to maintain an anaerobic environment. Yet, virtually nothing is known about oxygen levels in bladder urine even though bladder urine oxygen tension may both affect and be affected by the FUM.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Mueller, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brubaker L, Wolfe AJ. The new world of the urinary microbiota in women. Am J Obstet Gynecol. 2015 Nov;213(5):644-9. doi: 10.1016/j.ajog.2015.05.032. Epub 2015 May 21. PMID 26003055
- [Background] Pearce MM, Zilliox MJ, Rosenfeld AB, Thomas-White KJ, Richter HE, Nager CW, Visco AG, Nygaard IE, Barber MD, Schaffer J, Moalli P, Sung VW, Smith AL, Rogers R, Nolen TL, Wallace D, Meikle SF, Gai X, Wolfe AJ, Brubaker L; Pelvic Floor Disorders Network. The female urinary microbiome in urgency urinary incontinence. Am J Obstet Gynecol. 2015 Sep;213(3):347.e1-11. doi: 10.1016/j.ajog.2015.07.009. Epub 2015 Jul 23. PMID 26210757
- [Background] Brubaker L, Nager CW, Richter HE, Visco A, Nygaard I, Barber MD, Schaffer J, Meikle S, Wallace D, Shibata N, Wolfe AJ. Urinary bacteria in adult women with urgency urinary incontinence. Int Urogynecol J. 2014 Sep;25(9):1179-84. doi: 10.1007/s00192-013-2325-2. Epub 2014 Feb 11. PMID 24515544
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228